CLINICAL TRIAL: NCT01813578
Title: Effects of Intensive Aerobic and Muscle Endurance Exercise in Patients With Systemic Sclerosis - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Helene Alexanderson, PhD; RPT, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Norrbacka 2009; 0000 (Other Grant/Funding Number: Centre for care Science, KI, Norrbacka Eugeniastiftelsen)
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Exercise; Physical capacity; Aerobic capacity; Muscle function; Fatigue
MeSH Terms: conditions — Scleroderma, Systemic; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): An SSED study is an open-label design where the individual is his or her own control. All patients included received the same exercise intervention.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Intensive aerobic and muscle endurance exercise

SUMMARY:
The hypothesis is that intensive aerobic and endurance muscle training is safe and beneficial in patients with systemic sclerosis and concurrent interstitial lung disease.

The purpose of the study is to examine the effect of an eight week intensive aerobic exercise and muscle endurance training program for patients with systemic sclerosis and 50-100 % of forced vital capacity.

A single subject experimental design with repeated systematic measures during a six week A-phase (baseline period) and an eight week B-phase (intervention period) was used. Physical capacity (six minute walk test), aerobic capacity (submaximal treadmill test) and muscle endurance in shoulder and hip flexion (Functional Index 2) are assessed every other week throughout the 14 week study. Activity limitation (Health Assessment Questionnaire), quality of life (Short Form 36), Raynaud, Fatigue and Global Health during the recent week (Visual Analogue Scales) are assessed at weeks 0, 6, 14. The exercise program includes aerobic exercise corresponding to 15 on the Borg RPE scale (strenuous) and muscular endurance training three times/week.

DETAILED DESCRIPTION:
The purpose of the study is to examine the effect of an eight week intensive aerobic exercise and muscle endurance training program for patients with systemic sclerosis and 50-100 % of forced vital capacity.

As systemic sclerosis is a very rare condition a Single Subject Experimental Design (SSED) was used including a 6-week non-interventional A-phase where patients are assessed systematically followed by an 8-week interventional B-phase where patients exercise three days a week with continued systematic assessments. According to the 2-standard deviation (2 SD) band analysis, statistical analysis were performed for each patient individually. Accordingly, a statistically significant change was detected if two consecutive assessments in the B-phase exceeded the 2 standard deviations (SD) of the mean of the A-phase.

Patients were recruited from an ongoing study at the Karolinska University Hospital with the purpose to screen all patients with systemic sclerosis in Stockholm for cardiovascular disease. All patients meeting the inclusion criteria were invited to participate in this exercise study.

Assessments:

The six minute walking test was used to assess physical capacity. A submaximal treadmill test was used to estimate oxygen uptake in ml/kg x min. Muscle endurance was assessed by the Functional Index 2 registering the number of correct performed repetitions in 7 muscle groups. Pain, Raynaud's Phenomenon, fatigue and global disease impact on general well-being was assessed by the Visual Analogue scale (VAS), 0-100. Limitations in activities of daily living were assessed using the Health Assessment Questionnaire and the SF-36 was included to assess perceived health.

The Exercise program:

The program starts with a 10-minute warm-up session with biking at an intensity corresponding to perceived light exertion (10 on the Borg RPE, 6-20 scale). Thereafter, the load is increased to reach an intensity corresponding to perceived heavy exertion (15 on the Borg RPE scale) for an additional 15 minutes. During the last five minutes of the biking session, the loads are reduced to an intensity corresponding to light exertion. Heart rate was is recorded with a pulse watch (RS100 Polar) and peripheral saturation recorded with a heart rate oximeter (Wristox 3100 Nonin Medical). During the first weeks patients start on lower leads and increasing to the goal intensity. After the biking exercises, the participants perform repetitive dynamic muscle resistance training with the goal to achieve as many repetitions as possible in shoulder flexion and in hip flexion.

ELIGIBILITY:
Inclusion Criteria:

* limited or diffuse SSc
* age 18-80 years
* diagnosis duration > 1 year
* unchanged medication since 3 months
* 50-100 % of normal vital capacity
* exercising < once a week
* speak and understand the Swedish language
* average or below aerobic capacity according to the submaximal treadmill test (< 27 ml/kg x min for women and < 30 ml/kg x min for men)
* < 20 % reduced muscle endurance according to the Functional Index-2

Exclusion Criteria:

* Sendoxan treatment for alveolitis
* Pulmonal hypertension (PAH)
* heart condition contraindicating exercise
* < 50 % of normal vital capacity
* reduced kidney function
* not being able to perform the exercise program

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Six minute walking test assessing change in physical capacity compared to baseline. | At 0,2,4,6,8,10,12,14 weeks
  The six minute walking test assesses physical capacity by recording the walking distance achieved during 6 minutes. The participant is instructed to walk in a self-selected speed, but try to walk as fas a distance as possible. Heart rate, saturation and self-rated central and peripheral exertion is assessed at rest and after 2,4, and 6 minutes.

SECONDARY OUTCOMES:
Submaximal treadmill test. | Assessed at 0,2,4,6,8,10,12, and 14 weeks
  The Minor treadmill test assessed estimated oxygen uptake in ml/kg x min. The test requires a total of eight minutes where the first four minutes are performed on a horizontal treadmill with the patient walking at a self-elected walking speed. During the following four minutes, the patient continues at the same walking speed on a 5 % incline. Work heart rate, saturation, central and peripheral exertion according to the Borg RPE 6-20 scale were recorded after completion of the test.
Functional Index-2 | Assessed at 0,2,4,6,8,10,12 and 14 weeks.
  Functional Index 2 assessed muscle endurance by recording the number of correct performed repetitions in seven muscle groups; Shoulder flexion, shoulder abduction, neck flexion, hip flexion, knee extension, dorsal- and plantar flexion of the ankle. Maximal number of repetitions varies between 0-60 or 0-120 repetitions.

OTHER OUTCOMES:
Pain | Assessed at 0, 6 and 14 weeks
  Pain was rated on a Visual Analogue scale, 0-100
Raynaud's Phenomenon | Assessed at 0,6 and 14 weeks
  Patients rated impact of Raynaud's Phenomenon on a VAS, 0-00
Fatigue | Assessed at 0,6 and 14 weeks
  Patients rated fatigue on VAS, 0-100.
Disease impact on general well-being | Assessed at 0,6, and 14 weeks.
  Patients rated impact on well-being on a VAS, 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Alexanderson, PhD, RPT, Principal Investigator — Karolinska University Hospital / Karolinska Institutet
Locations (1):
- Karolinska Univeristy Hospital, Solna, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Alexanderson H, Bergegard J, Bjornadal L, Nordin A. Intensive aerobic and muscle endurance exercise in patients with systemic sclerosis: a pilot study. BMC Res Notes. 2014 Feb 7;7:86. doi: 10.1186/1756-0500-7-86. PMID 24507585